CLINICAL TRIAL: NCT01105143
Title: Effects of Negative Energy Balance on Muscle Mass Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Professor Joachim Spranger, Professor, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA 20100415
Record Dates: First submitted 2010-04-14; First posted 2010-04-16 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Weight Loss; Obesity; Skeletal Muscle; Insulin Sensitivity/Resistance
Keywords: weight loss; muscle mass
MeSH Terms: conditions — Weight Loss; Obesity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- lifestyle intervention (Active Comparator): Multimodal lifestyle intervention to reduce body weight
  Interventions: Behavioral: multimodal lifestyle intervention
- placebo (Placebo Comparator): placebo
  Interventions: Behavioral: placebo

INTERVENTIONS:
Behavioral: multimodal lifestyle intervention — multimodal lifestyle intervention will be performed to reduce body weight
  Arms: lifestyle intervention
Behavioral: placebo — no intervention, only follow up
  Arms: placebo

SUMMARY:
The investigators here propose to perform a prospective randomized intervention trial in post-menopausal women to investigate the endocrine network, which contributes to the changes in skeletal muscle mass during weight loss.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 27 kg/m2 (adults)
* postmenopausal state

Exclusion criteria:

* weight loss of more than 5kg in the last 2 months x
* unhealthy patients with: severe chronic diseases including cancer within the last 5 years, severe heart disease, severe impairment of hepatic or renal function, severe anaemia or disturbed coagulation
* eating disorders or any other psychiatric condition that would interact with the trial intervention
* malabsorption
* acute or chronic infections
* severe hypertension
* myopathy
* food allergies
* any other uncontrolled endocrine disorder
* changes of smoking habits, diets or medication that strongly affects energy homeostasis within the last 3 months prior to study inclusion

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Changes of myocellular insulin sensitivity (hyperinsulinemic clamp) during negative energy balance and during stabilized modification of body composition after weight loss. | 4 months
  Analysis of myocellular insulin sensitivity by hyperinsulinemic clamp in mg•kg-1•min-1/(mU•L-1)
Changes of skeletal muscle mass (air displacement plethysmography) during negative energy balance and during stabilized modification of body composition after weight loss. | 4 months
  Analysis of muscle mass (in % of body weight)

SECONDARY OUTCOMES:
Effects on energy expenditure | 4 months
  Measurement of energy expenditure (kcal/d), postprandial thermogenesis (%) and respiratory coefficient
Effects on myocellular and adipose tissue metabolism and substrate utilization | 4 months
  Measurement of myocellular and adipose metabolism using microdialysis (glycerol (µmol/l), lactate (mmol/l), pyruvate (µmol/l), glucose (mmol/l)) during oral glucose load (180 minutes)
Effects on myocellular and adipose tissue mRNA expression | 4 months
  Analysis of myocellular and adipose mRNA expression (RNA sequencing) in counts
Weight regain | 24 months
  Analysis of body weight regain (BMI; kg/m2) during follow up
Fat mass | 24 months
  Analysis of body fat (kg and %)
Measurement of human gut microbiome at baseline, during weight loos, after weight loss (negative energy balance) and during stabilized modification of body composition 4 weeks after weight loss | 4 months
  16S rRNA sequencing and/or shotgun metagenomic pyrosequencing of the gut microbiota for assessment of microbiota composition and gene abundances.

OTHER OUTCOMES:
FFA during negative energy balance and during stabilized modification of body composition after weight loss. | 12 months
  Measurement of fatty acids at baseline, during negative energy balance, during stabilized modification of body composition after weight loss and during follow up.
Metanephrines during negative energy balance and during stabilized modification of body composition after weight loss. | 12 months
  Measurement of metanephrines at baseline, during negative energy balance, during stabilized modification of body composition after weight loss and during follow up.
Leptin during negative energy balance and during stabilized modification of body composition after weight loss. | 12 months
  Measurement of leptin at baseline, during negative energy balance, during stabilized modification of body composition after weight loss and during follow up.
Cortisol during negative energy balance and during stabilized modification of body composition after weight loss. | 12 months
  Measurement of cortisol at baseline, during negative energy balance, during stabilized modification of body composition after weight loss and during follow up.
Follistatin during negative energy balance and during stabilized modification of body composition after weight loss. | 12 months
  Measurement of follistatin at baseline, during negative energy balance, during stabilized modification of body composition after weight loss and during follow up.
Adiponectin during negative energy balance and during stabilized modification of body composition after weight loss. | 12 months
  Measurement adiponectin at baseline, during negative energy balance, during stabilized modification of body composition after weight loss and during follow up.
Natriuretic peptide during negative energy balance and during stabilized modification of body composition after weight loss. | 12 months
  Measurement of natriuretic peptide at baseline, during negative energy balance, during stabilized modification of body composition after weight loss and during follow up.
IGF-1 during negative energy balance and during stabilized modification of body composition after weight loss. | 12 months
  Measurement of IGF-1 at baseline, during negative energy balance, during stabilized modification of body composition after weight loss and during follow up.
Analysis of predictive impact of several hormonal and metabolic parameters on body weight regain, course of insulin sensitivity and metabolism | 24 months
  The effect of measured parameters (see other endpoints) on long-term course of BMI, muscle mass, insulin sensitivity and energy expenditure will be analyzed using mathematical models

CONTACTS AND LOCATIONS:
Overall Officials: Knut Mai, Prof, Principal Investigator — Charite
Locations (1):
- Charite, Berlin, Germany

REFERENCES:
- [Derived] Spranger L, Weiner J, Bredow J, Zeitz U, Grittner U, Boschmann M, Dickmann S, Stobaus N, Schwartzenberg RJ, Brachs M, Spranger J, Mai K. Thrifty energy phenotype predicts weight regain in postmenopausal women with overweight or obesity and is related to FGFR1 signaling. Clin Nutr. 2023 Apr;42(4):559-567. doi: 10.1016/j.clnu.2023.02.020. Epub 2023 Feb 24. PMID 36863292
- [Derived] Sbierski-Kind J, Grenkowitz S, Schlickeiser S, Sandforth A, Friedrich M, Kunkel D, Glauben R, Brachs S, Mai K, Thurmer A, Radonic A, Drechsel O, Turnbaugh PJ, Bisanz JE, Volk HD, Spranger J, von Schwartzenberg RJ. Effects of caloric restriction on the gut microbiome are linked with immune senescence. Microbiome. 2022 Apr 4;10(1):57. doi: 10.1186/s40168-022-01249-4. PMID 35379337
- [Derived] Koppel N, Bisanz JE, Pandelia ME, Turnbaugh PJ, Balskus EP. Discovery and characterization of a prevalent human gut bacterial enzyme sufficient for the inactivation of a family of plant toxins. Elife. 2018 May 15;7:e33953. doi: 10.7554/eLife.33953. PMID 29761785